CLINICAL TRIAL: NCT04022785
Title: A Phase I Study of PLX51107 (A Novel Bromodomain Inhibitor) in Combination With Azacytidine for Patients With Myelodysplastic Syndrome and Acute Myeloid Leukemia (AML)
Brief Title: PLX51107 and Azacitidine in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0725; NCI-2019-02517 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0725 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Myelodysplastic/Myeloproliferative Neoplasm; Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Myeloproliferative Disorders | interventions — Azacitidine; PLX51107

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (BRD4 Inhibitor PLX51107, azacitidine) (Experimental): Patients receive PLX51107 PO QD on days 1-21 and azacitidine SC or IV over 15 minutes on days 8-14 and 22-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: BRD4 Inhibitor PLX51107

INTERVENTIONS:
Drug: Azacitidine — Given IV or SC
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: BRD4 Inhibitor PLX51107 — Given PO
  Other Names: PLX 51107; PLX-51107; PLX51107

SUMMARY:
This phase I trial studies the side effects and best dose of PLX51107 and how well it works with azacitidine in treating patients with acute myeloid leukemia or myelodysplastic syndrome. PLX51107 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving PLX51107 and azacitidine may work better than azacitidine alone in treating patients with acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the minimum safe and biologically-effective dose of the combination of PLX51107 and azacitidine (AZA).

SECONDARY OBJECTIVES:

I. To determine overall response rate (ORR) rate including CR (complete remission) + CRp (complete remission with incomplete platelet recovery) + CRi (complete remission with incomplete count recovery) + CRh (complete remission with partial hematologic recovery), partial remission (PR) within 3 months of treatment initiation of PLX51107 and AZA combination in patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

II. To investigate correlations of response to this combination with a pre-therapy, on-therapy, and progression 81-gene panel of gene mutations in AML.

III. To determine the duration of response (DOR), event-free survival (EFS), overall survival (OS), and number of patients bridged to stem cell transplant (SCT) and median duration to SCT from the initiation of the combination.

OUTLINE: This is a dose-escalation study of PLX51107.

Patients receive PLX51107 orally (PO) once daily (QD) on days 1-21 and azacitidine subcutaneously (SC) or intravenously (IV) over 15 minutes on days 8-14 and 22-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 6-12 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of

  * AML (World Health Organization [WHO] classification definition of >= 20% blasts), or
  * MDS intermediate-2 score or with > 10% blasts, to include: MDS, myeloproliferative neoplasm (MPN) with 10% blasts or more, or MDS/MPN 10% blasts or more
* Patients who have received at least one prior therapy for AML or for MDS will be eligible. Any prior therapy for AML or MDS will be counted as a prior salvage
* In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of protocol therapy will be at least 2 weeks for cytotoxic agents or at least 5 half-lives for cytotoxic/non-cytotoxic agents. The half-life for the therapy in question will be based on published pharmacokinetic literature (abstracts, manuscripts, investigator brochures, or drug-administration manuals) and will be documented in the protocol eligibility document. The use of chemotherapeutic or anti-leukemic agents is not permitted during the study with the following exceptions:

  * Intrathecal (IT) therapy for patients with controlled central nervous system (CNS) leukemia at the discretion of the principal investigator (PI). Controlled CNS leukemia is defined by the absence of active clinical signs of CNS disease and no evidence of CNS leukemia on the most recent 2 simultaneous cerebrospinal fluid (CSF) evaluations
  * Use of one dose of cytarabine (up to 2 g/m^2) or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first four weeks on therapy. These medications will be recorded in the case-report form.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measured or calculated creatinine clearance >= 60 mL/min (unless considered due to leukemia)
* Total bilirubin < 1.8 mg/dL (unless increase is due to hemolysis, congenital disorder, or leukemia)
* Transaminases (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x upper limit of normal (ULN) (unless considered due to leukemia)
* Potassium levels should be within institutional normal limits (unless considered due to leukemia)
* Magnesium levels should be within institutional normal limits (unless considered due to leukemia)
* Calcium (normalized for albumin) levels should be within institutional normal limits (unless considered due to leukemia)
* Ability to take oral medication
* Ability to understand and provide signed informed consent prior to any study-related procedures and to comply with all study requirements
* Baseline left ventricular ejection fraction by echocardiogram (ECHO) or multigated acquisition scan (MUGA) >= 50%
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 7 days. Men must agree not to father a child and agree to use a condom if his partner is of child bearing potential
* WOCBP must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy until after the last dose of investigational drug. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as men with azoospermia do not require contraception

Exclusion Criteria:

* Patients with known significant impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PLX51107
* Patients with any other known concurrent severe and/or uncontrolled medical condition including but not limited to diabetes, cardiovascular disease including hypertension, renal disease, or active uncontrolled infection, which could compromise participation in the study. Patients on active antineoplastic or radiation therapy for a concurrent malignancy at the time of screening. Maintenance therapy, hormonal therapy, or steroid therapy for well-controlled malignancy is allowed
* Patients with known positive human immunodeficiency virus (HIV), hepatitis B or C infection by serology, with the exception of those with an undetectable viral load within 3 months. (HIV testing and hepatitis B or C testing is not required prior to study entry). Subjects with serologic evidence of prior vaccination to hepatitis B virus (HBV) (i.e., hepatitis B virus surface antigen negative [HBs Ag-], and hepatitis B surface antibody positive [HBs+]) may participate
* Patients with advanced malignant hepatic tumors
* Patients with known hypersensitivity to AZA or mannitol
* Women who are pregnant or are breast-feeding
* Patients who receive strong CYP3A4 and CYP2C8 inhibitors or inducers or CYP3A4 substrate drugs with a narrow therapeutic range, taken within 14 days or 5 drug half-lives, whichever is longer, before start of study drug
* Patients who have received anti-cancer therapy within 14 days (or 5 half-lives) with all toxicities resolved to grade 1 or less. No immune therapy or other biologic therapy (other monoclonal antibodies or antibody-drug conjugates [ADCs]) within 28 days of cycle 1 day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Toxicity type and severity will be summarized for each patient cohort using frequency tables. Per-treated analysis will be performed to include any patient who received the treatment regardless of the eligibility nor the duration or dose of the treatment received.
Minimum safe and biologically effective dose | Up to 28 days
  The minimum safe and biologically-effective dose is the highest dose level in which < 2 patients of 6 develop first cycle dose limiting toxicity.

SECONDARY OUTCOMES:
Overall response rate | Within 3 months of treatment initiation
  Will be defined as blast count reduction, hematologic improvement, partial remission, complete remission (CR), complete remission with incomplete count recovery, complete remission with incomplete platelet recovery, complete remission with partial hematologic recovery. Will be calculated and credible interval will be provided. Wilcoxon rank sum test or Fisher's exact test will be used to evaluate the association between patient prognostic factor (e.g. lab result and gene mutation) and response.
Gene mutations in acute myeloid leukemia | Up to 5 years
  Pre-therapy, on-therapy, and progression 81-gene panel of gene mutations will be correlated with response.
Duration of response | Number of days from the date of initial response to the date of first documented disease progression/relapse or death, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Event-free survival | Number of days from the date of treatment initiation to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Overall survival | Time from treatment start until death or last follow up, assessed up to 5 years
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Number of patients bridged to stem cell transplant (SCT) | Up to 5 years
Median duration to SCT from initiation of combination | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Pemmaraju, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org